CLINICAL TRIAL: NCT07276165
Title: Reliability and Validity of the Turkish Version of the Adolescent Idiopathic Scoliosis-Truncal Anterior Asymmetry Scoliosis Questionnaire (TAASQ)
Brief Title: Reliability and Validity of the Adolescent Idiopathic Scoliosis - Truncal Anterior Asymmetry Scoliosis Questionnaire (TAASQ)
Status: Not yet recruiting | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assist. Prof. Dr., Hasan Kalyoncu University
Other Study IDs: 2024/49
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Idiopathic Adolescent; Scoliosis Define Themselves; Physical Perception of Their Bodies
Keywords: Scoliosis; Body appearance; Female
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scoliosis Group: The study sample consists of female individuals between the ages of 10-18 diagnosed with adolescent idiopathic scoliosis.

SUMMARY:
The survey examines how individuals with scoliosis define themselves and their physical appearance. Our aim in this study was to translate this survey into Turkish and demonstrate its reliability and validity.

DETAILED DESCRIPTION:
The "Adolescent Idiopathic Scoliosis-Truncal Anterior Asymmetry Scoliosis Questionnaire" was developed to investigate how individuals with scoliosis feel about their frontal body appearance. The survey was developed by BS Lonner and colleagues and published in 2023. It consists of 14 questions. Female patients with scoliosis are asked to answer these questions personally. Permission for the Turkish validity and reliability of the survey was requested and received on November 18, 2024. The survey questions how individuals with scoliosis define themselves and their physical perception of their bodies. The aim of this study is to translate this survey into Turkish and demonstrate its reliability and validity. This study will examine the test-retest reliability and internal consistency of the Adolescent Idiopathic Scoliosis-Truncal Anterior Asymmetry Scoliosis Questionnaire (TAASQ), and its validity with the SRS-22 and Walter Reed questionnaires. This study was designed as an intra-rater and intra-rater reliability and structural validity study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent idiopathic diagnosis

Exclusion Criteria:

* Individuals who did not agree to participate in the study

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female individuals diagnosed with adolescent idiopathic scoliosis between the ages of 10-18 will be evaluated within the scope of the study.
Study Population: The sample group consisted of female adolescents with idiopathic scoliosis who volunteered for the study and met the inclusion criteria. Convenience sampling was used in sample selection.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Adolescent Idiopathic Scoliosis-Truncal Anterior Asymmetry Scoliosis Questionnaire (TAASQ) | through of the study, average 4 months
  The "Adolescent Idiopathic Scoliosis-Truncal Anterior Asymmetry Scoliosis Questionnaire" was developed to ask individuals with scoliosis how they feel about the frontal appearance of their bodies. The survey was developed by BS Lonner and colleagues and published in 2023. The survey consists of 14 questions. Female patients with scoliosis are asked to answer these questions themselves.A high score indicates poor body appearance.

SECONDARY OUTCOMES:
Scoliosis Research Society-22 (SRS-22) | through of the study, average 4 months
  The SRS-22 questionnaire includes five domains. The domains and the number of questions in them are as follows: function/activity (5), pain (5), self-image/appearance (5), mental health (5), and satisfaction with management (2). The combination of the first 4 domains is labeled subtotal. The mental health questions are adapted with permission from SF-36. The scoring scale ranges from 5 as best to 1 as worst.
Walter Reed Visual Assessment Scale | through of the study, average 4 months
  The Walter Reed Visual Assessment Scale (WRGDS) was developed by Pineda et al. in 2006 to measure the perceived severity of deformity in individuals with scoliosis, using visual patterns. The scale assesses spinal deformity, rib protrusion, lumbar protrusion, thoracic deformity, trunk imbalance, scapular asymmetry, and shoulder asymmetry. In each section, the individual is asked to mark the image closest to their own image from five different visuals representing the degree of deformity. Scoring is performed with a score of 1 representing the image with minimal deformity and a score of 5 representing the image with maximum deformity. A high score indicates a high perceived deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba GÖNEN, Asisst. Prof. Dr., Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alanay A, Cil A, Berk H, Acaroglu RE, Yazici M, Akcali O, Kosay C, Genc Y, Surat A. Reliability and validity of adapted Turkish Version of Scoliosis Research Society-22 (SRS-22) questionnaire. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2464-8. doi: 10.1097/01.brs.0000184366.71761.84. PMID 16261127
- [Result] Asher M, Min Lai S, Burton D, Manna B. The reliability and concurrent validity of the scoliosis research society-22 patient questionnaire for idiopathic scoliosis. Spine (Phila Pa 1976). 2003 Jan 1;28(1):63-9. doi: 10.1097/00007632-200301010-00015. PMID 12544958
- [Result] Sanders JO, Polly DW Jr, Cats-Baril W, Jones J, Lenke LG, O'Brien MF, Stephens Richards B, Sucato DJ; AIS Section of the Spinal Deformity Study Group. Analysis of patient and parent assessment of deformity in idiopathic scoliosis using the Walter Reed Visual Assessment Scale. Spine (Phila Pa 1976). 2003 Sep 15;28(18):2158-63. doi: 10.1097/01.BRS.0000084629.97042.0B. PMID 14501929
- [Result] Alhada TL, Castel LC, Pfirrmann C, Davoust L, Loot M, Angelliaume A, Harper L, Lefevre Y. Translation and validation of the French version of the adolescent idiopathic scoliosis Truncal Anterior Asymmetry Scoliosis Questionnaire (TAASQ). Spine Deform. 2023 Nov;11(6):1363-1369. doi: 10.1007/s43390-023-00736-4. Epub 2023 Aug 2. PMID 37531015